CLINICAL TRIAL: NCT02927730
Title: The Correlation Between Clinical Diagnosis of Retained Placenta And Histology
Acronym: WHI
Status: Completed | Type: Observational
Sponsor: Bait Balev Hospital (Other)
Collaborators: Maccabi Healthcare Services, Israel (Other)
Responsible Party: Sponsor
Other Study IDs: BaitBHresiduaCTIL
Record Dates: First submitted 2016-10-06; First posted 2016-10-07 (Estimated); Last update posted 2020-02-05 (Actual); Status verified 2016-09

CONDITIONS: Retained Product of Pregnancy
Keywords: Retained placenta, surgical hysteroscopy, residua
MeSH Terms: conditions — Placenta, Retained

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- positive retainted placenta histology: base on chorionic villi in the pathalogic sample
  Interventions: Other: no interventions
- negative retainted placenta histology
  Interventions: Other: no interventions

INTERVENTIONS:
Other: no interventions — no interventions

SUMMARY:
The main purpose is to evaluate the correlation in qualitative and quantitative manner between clinical diagnosis of retained placenta and histology. Secondly, to assess different clinical parameters that are likely related to accuracy of the diagnosis of RPOC

DETAILED DESCRIPTION:
Background:

Retained products of conception (RPOC) are a common and treatable complication after delivery or termination of pregnancy. The reported incidence in the literature is around 1% of all pregnancies. Most often, diagnoses are made on clinical basis and there is only scarce information available related to the correlation between the clinical and pathological diagnosis of RPOC. The gold standard for diagnosis of RPOC is based on histopathological confirmation of chorionic villi in tissue derived from the uterus. Once RPOC is diagnosed on a clinical basis, several treatment options are available, including expectant management, pharmacological treatment, and surgical interventions. Given the risks associated with surgical interventions, accurate diagnosis is vital. Guidelines at Maccabi Health Care Organization mandate that hysteroscopic removal of suspected RPOC should be performed only after approval by a Gynecological Surgical Preauthorization committee. Based on the activity of this committee and starting 2011, Maccabi has developed a database on certain gynecologic-surgical procedures including hysteroscopic removal of suspected RPOC.

Purpose of the study:

The main purpose is to evaluate the correlation in qualitative and quantitative manner between clinical diagnosis of retained placenta and histology.

Expected results:

70% correlation between the clinical and pathological diagnosis of RPOC.

Methods:

Establishing a dedicated database which includes demographic, clinical and histological data of women who have undergone hysteroscopic removal of suspected RPOC and statistical assessment of correlations.

Significance:

Determination of the correlation between clinical suspicion and histological diagnosis of retained placental tissue Finding clinical parameters that may increase the accuracy of this diagnosis and will help to prevent unnecessary procedures.

ELIGIBILITY:
Inclusion Criteria:

* Women who diagnosed clinically with RPOC
* women who prefomed therapeutic hysteroscopy under the diagnosis of RPOC

Exclusion Criteria:

* Women who underwent hysteroscopy presumptive diagnosis of RPOC without documentation of pathological results were excluded.
* Women who have not performed / recorded sonography test before the hysterocpy.

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Study population consists of women who were diagnosed clinically with the rest of the placenta after birth or termination of pregnancy (miscarriage or artificial). The women passed the approval of the Commission and undergo therapeutic hysteroscopy. The information is taken from a database of relevant actions Maccabi Healthcare Services, and includes data from 2012 to 2015.
Sampling Method: Probability Sample
Enrollment: 240 (Actual)
Dates: Start 2016-09; Primary Completion 2016-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
the correlation between clinical suspicion and histological diagnosis of retained placental tissue Finding is 67.5 %. | sep-oct 2016

SECONDARY OUTCOMES:
No clinical symptoms increase the accuracy of this diagnosis. There no advantage in the use of diagnostic hysteroscopy in case of suspected retainted placenta. | sep-oct 2016